CLINICAL TRIAL: NCT05911503
Title: A Clinical Study of High Concentration(2%) Ganciclovir Eye Drops in the Treatment of Cytomegalovirus Retinitis
Brief Title: Clinical Study of High Concentration Ganciclovir Eye Drops in the Treatment of Cytomegalovirus Retinitis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Principal Investigator,MD,PhD, Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023KY-23
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Cytomegalovirus Retinitis; Ganciclovir Eye Drops
MeSH Terms: conditions — Cytomegalovirus Retinitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2% Ganciclovir Eye Drops therapy Group (Experimental): Administration method and dosage adjustment: 2% ganciclovir eye drops, 10 times/day for two weeks, 8 times/day for two weeks, 6 times/day for two weeks, 4 times/day for more than 6 weeks
  Interventions: Drug: 2% Ganciclovir Eye Drops

INTERVENTIONS:
Drug: 2% Ganciclovir Eye Drops — Administration method and dosage adjustment: 2% ganciclovir eye drops, 10 times/day for two weeks, 8 times/day for two weeks, 6 times/day for two weeks, 4 times/day for more than 6 weeks

SUMMARY:
Clinical study of high concentration ganciclovir eye drops in the treatment of cytomegalovirus retinitis

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the use of 2% Ganciclovir Eye Drops, its potential risks and benefits. This is a monocencer, single arm, prospective study. The experimental group is: 2% Ganciclovir Eye Drops therapy group.

Administration method and dose adjustment: 2% ganciclovir eye drops, 10 times / day for two weeks, 8 times/day for two weeks, 6 times/day for two weeks, 4 times/day for more than six weeks.

According to best corrected visual acuity (BCVA), intraocular pressure, corneal abrasion, anterior chamber and vitreous inflammation, optical coherence tomography (OCT), Ultra wide angle fundus image and so on. The investigators evaluate the effects of 2% Ganciclovir Eye Drops in treatment of cytomegalovirus retinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in studies and sign informed consent forms
2. Ages 2-80 years (with cut-off values) male and female
3. One of the following is true （1）In patients with cytomegalovirus retinitis after hematopoietic stem cell transplantation/cord blood transplantation, the white blood cell count is less than 4× 10^9/L, and the platelet count ranges are 25× 10^9/L≤ PLT<100×10^9/L，Intravitreal injection carries a greater risk of infection and bleeding, and is unable to administer systemic medication due to the bone marrow suppression of antiviral drugs, or systemic medication for severe CMV retinitis cannot be well controlled; （2）In patients with CMVR with AIDS, the CD4+ T cell count is less than 100/μl, there is a great risk of infection with intravitreal injection, and the systemic medication of severe CMV retinitis cannot be well controlled.

Exclusion Criteria:

* Eye condition

  1. The presence of refractive interstitial opacification affects fundus observation;
  2. Intravitreal ganciclovir or sodium phosformate injections were performed within 1 week prior to baseline;
  3. Other diseases that can affect visual function such as syphilis-related eye diseases, acute retinal necrosis, congenital glaucoma, congenital corneal lesions, congenital macular degeneration, etc.
* General condition

  1. Severe neutropenia (<0.5×10^9) or severe thrombocytopenia (< 25× 10^9/L);
  2. Other investigators judged patients who were not suitable for enrollment;

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Fundus lesions | 24 weeks
  The size changes of fundus lesions after medication are recorded

SECONDARY OUTCOMES:
Change In LogMAR Best Corrected Visual Acuity (BCVA)From Baseline to Each visit | 24 weeks
  The size changes of fundus lesions after medication are recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided